CLINICAL TRIAL: NCT03690518
Title: Impact of Cardiovascular Rehabilitation on the Quality of Life of Adolescents and Young Adults With Congenital Heart Disease: A Randomized Controlled Multicentre Trial
Brief Title: Rehabilitation of Adolescents and Young Adults With Congenital Heart Diseases
Acronym: QUALIREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0039; 7576 (Other: UH Montpellier)
Record Dates: First submitted 2018-08-07; First posted 2018-10-01 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Heart Defects, Congenital; Adolescent; Young Adult
Keywords: cardiac rehabilitation; Congenital heart diseases; Heart defects, congenital; Adolescent; Young adult; Physical activity; Cardio-pulmonary exercice test; Oxygen uptake; Muscular deconditioning; Patient education as topic; Quality of life; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity; Behavior | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Cardiac rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Controls will have a regular follow-up without any intervention (no rehabilitation program)
- Rehabilitaiton (Active Comparator): Cardiac rehabilitation: Rehabilitation will have a regular follow-up with intervention (rehabilitation program)
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — Educational/Counseling/Training : Rehabilitation, , cardiovascular rehabilitation in congenital heart disease
  Arms: Rehabilitaiton

SUMMARY:
The investigators aim to measure the impact of a rehabilitation program in congenital cardiology in terms of health related quality of life. The orginality of the rehabilitation program consists in its design : initial hospitalizationfor a short period of time (5 days) at the rehabilitation center, followed by 11 weeks of rehabilitation at home under the supervision of a specialized sports trainer.

DETAILED DESCRIPTION:
Adolescents and adults with congenital heart disease (CHD) have reduced exercise capacity compared to the general population, even for "simple" heart disease.

Regular physical activity is known to reduce the risk of acquired heart disease.

Cardiac rehabilitation programs have been largely developed to manage adult coronary and heart failure patients, which is not yet the case routinely in patients, adults and children, carriers of DC.

The investigators assume that patients who participate in this program will improve their quality of life compared to controls.

The orginality of the rehabilitation program consists in its design : initial hospitalizationfor a short period of time (5 days) at the rehabilitation center, followed by 11 weeks of rehabilitation at home under the supervision of a specialized sports trainer .

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 13 to 25 years included
* With a congenital heart diseases (CHD) as defined in the international CHD classification.
* Recent (< 3 months) cardio-pulmonary exercise test (CPET)with maximum oxygen uptake (VO2max) <80% of theoretical values and/or first ventilatory anaerovic threshold (VAT) <55% of VO2max.
* Consent of the adult patient or the parents or legal guardians of the minor patient.
* Beneficiary of the social security scheme.

Exclusion Criteria:

* Uncontrolled arrhythmia.
* Cardiac surgery planned during the rehabilitation program.
* Severe musculoskeletal disorders.
* Severe intellectual disability that does not allow the quality of life questionnaire to be completed.
* Pregnancy.
* Patient who already underwent cardiac rehabilitation in the last 24 months.
* All medical contraindications to perform a cardiorespiratory stress test.
* Uncontrolled heart failure (NYHA IV)
* Obesity (BMI > 30)

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Quality of life score (PedsQL, 24 items), range score from 0 to 100, higher score indicating better quality of life. | follow up of patients over 12 months
  Evolution of the PedsQL 4.0 self-reported scores from month 0 to month 12

SECONDARY OUTCOMES:
Peak oxygen uptake (VO2max, ml/kg/min) | Month 0 and Month 12
ventilatory anaerobic threshold (VAT, ml/kg/min) | Month 0 and Month 12
knowledge of the disease | Month 0 and Month 12
  Disease knowledge questionnaire (Leuven questionnaire, 34 items, total range score from 0 to 100, a higher score indicating better knowledge)
cardiac events | Month 0 and Month 12
  number of consultation in cardiology, number of hospitalization in cardiology, number of cardiovascular events
physical activity scoring | Month 0 and Month 12
  Score of physical activity (Ricci and Gagnon questionnaire, 9 items, total range score from 6 to 45, higher score indicating a higher level of physical activity)
functional NYHA class | Month 0 and Month 12
  NYHA functional class= New York Association functional class from the World Health Organization
Cardiac output during exercise | Month 0 and Month12
  Variation of cardiac output during exercise tests measured by impedance measurement (Physioflow)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Haut Lévêques - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Gabriel Montpied Hospital- Clermont Ferrand University Hospital, Clermont-Ferrand
  - Grenoble Alpes University Hospital, Grenoble
  - Marie Lannelongue Hospital, Le Plessis-Robinson
  - Children and Mother Hospital - Limoges University Hospital, Limoges
  - La Timone- Public Assistance - Marseille hospitals, Marseille
  - Liberal Cabinet Massy, Massy
  - Arnaud de Villeneuve - University Hospital, Montpellier
  - Nice University Hospital, Nice
  - Caremeau - Nimes University Hospital, Nîmes
  - Saint-Pierre Institute, Palavas-les-Flots
  - Necker - Sick Children Hospital - Paris, Paris
  - La Miletrie -Poitier University Hospital, Poitiers
  - Children Hospital - Toulouse University Hospital, Toulouse
  - Pasteur Clinic, Toulouse
  - Barbois Hospital - Nancy University Hospital, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Amedro P, Gavotto A, Legendre A, Lavastre K, Bredy C, De La Villeon G, Matecki S, Vandenberghe D, Ladeveze M, Bajolle F, Bosser G, Bouvaist H, Brosset P, Cohen L, Cohen S, Corone S, Dauphin C, Dulac Y, Hascoet S, Iriart X, Ladouceur M, Mace L, Neagu OA, Ovaert C, Picot MC, Poirette L, Sidney F, Soullier C, Thambo JB, Combes N, Bonnet D, Guillaumont S. Impact of a centre and home-based cardiac rehabilitation program on the quality of life of teenagers and young adults with congenital heart disease: The QUALI-REHAB study rationale, design and methods. Int J Cardiol. 2019 May 15;283:112-118. doi: 10.1016/j.ijcard.2018.12.050. Epub 2018 Dec 20. PMID 30616811